CLINICAL TRIAL: NCT00692445
Title: A Multi-Center, Double Blind, Randomized, Placebo-Controlled, Parallel Group, Flexible Dose Titration, Add-On Study of TC-5214 in the Treatment of MDD With Subjects Who Are Partial Responders or Non-Responders to Citalopram Therapy
Brief Title: TC-5214 as add-on the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TC-5214-23-CRD-001
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Major Depressive Disorder; Depression
Keywords: depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Citalopram; Mecamylamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- citalopram + TC-5214 (Active Comparator)
  Interventions: Drug: TC-5214 + citalopram
- citalopram + placebo (Placebo Comparator)
  Interventions: Drug: Placebo + citalopram

INTERVENTIONS:
Drug: TC-5214 + citalopram — TC-5214 (as TC-5214-23) will be provided as white, opaque, hard-gelatin capsules in strengths of 1, 2, and 4 mg.
  Other Names: Mecamylamine
  Arms: citalopram + TC-5214
Drug: Placebo + citalopram — Placebo will be provided with exactly the same shape, size and appearance. Subjects will take 2, 4, or 8 mg of study drug (or matching placebo), divided BID.
  Other Names: Placebo; Citalopram
  Arms: citalopram + placebo

SUMMARY:
This is a multi-center, double blind, randomized, placebo-controlled, parallel group, flexible dose titration study conducted in centers in the USA and India. Following a washout period, subject will be treated with citalopram 20 mg once daily for 4 weeks, then with 40 mg once daily for 4 weeks. Subjects who tolerate 40 mg citalopram, but whose MADRS score is < 50% from baseline, but no lower than 17, will be considered partial or non-responders and will be randomized to receive either placebo or TC-5214 as add-on therapy. TC-5214 or placebo will be started at 2 mg daily (BID dosing), and be titrated based on tolerability and therapeutic response up to 8 mg daily. Approximately 560 subjects will enter the Open Label Phase and approximately 220 will enter the double blind phase of the study.

DETAILED DESCRIPTION:
This is a multi-center, double blind, randomized, placebo-controlled, parallel group, flexible dose titration study conducted in centers in the USA and India.

Following a washout period, subject will be treated with citalopram 20 mg once daily for 4 weeks, then with 40 mg once daily for 4 weeks. Subjects who tolerate 40 mg citalopram, but whose MADRS score is reduced 50% from baseline, but no lower than 17, will be considered partial or non-responders and will be randomized to receive either placebo or TC-5214 as Add:-on therapy.

TC-5214 or placebo will be started at 2 mg daily (1mg BID dosing). After 2 weeks treatment, medication can be increased to 4 mg (2mg BID) or continued unchanged. Dose escalation will depend on good tolerability and inadequate therapeutic response. After a further 2 weeks, medication can be increased to 8 mg (4mg BID) if felt appropriate by the investigator. Again, dose escalation will depend on good tolerability and inadequate therapeutic response. At any time during the double blind phase of the study, placebo or TC-5214 can be reduced to the last previous dose level following the emergence of unacceptable adverse event(s).

If a subject is prematurely discontinued from the study between Week 8 and Week 16 for any reason, the investigator will make every effort to perform all evaluations as per protocol, assuming the subject had reached the end of the double blind Add:-on treatment phase. These evaluations are to be made as soon as possible but within 2 weeks of discontinuation.

For the subjects completing the double blind phase of the study, there will be a follow-up visit 2-3 weeks after the last dose of trial medication. At this follow-up, any signs or symptoms of relapse will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of major depressive disorder (MDD) according to DSM-IV and confirmed via MINI diagnostic scale
2. No more than 1 prior antidepressant course of treatment before trial entry.
3. Able to give written informed consent.
4. MADRS score greater than 27.
5. CGI-S score greater than or equal to 4.
6. No clinically significant abnormality on physical examination, vital signs, ECG or laboratory tests at screening.
7. Women of child bearing potential must: a) have a negative urine pregnancy test, b) not be nursing, and c) be willing to use acceptable methods of contraception throughout the study period.

Exclusion Criteria:

1. Any co morbid psychiatric illness confirmed by MINI diagnostic scale, especially bipolar disorder, schizophrenia, dementia, or PTSD
2. Subjects with significant suicidal risk upon clinical assessment utilizing the M.I.N.I.
3. History of alcohol or drug abuse over the last 6 months
4. History of seizures or seizure disorders
5. Any other severe progressive and uncontrolled medical condition
6. For other controlled medical conditions, medication to be unchanged over the 2 months preceding screening, or else the subject will be excluded
7. Subjects with Glaucoma, Kidney Disease or Heart Disease
8. Known hypersensitivity to mecamylamine
9. Other investigational drug in previous 30 days
10. Screening QTcB or QTcF > 450 msec
11. Current or prior citalopram treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Mean change between TC-5214 and placebo from DB baseline (Week 8) of the HAMD-17 score, at Week 16. | 16 Weeks

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 16 Weeks
  Treatment emergent adverse events (TEAEs) will be tabulated and summarized by presenting the incidence (number of subjects) in each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo N Rivera, MD, Principal Investigator — Community Research
Locations (27):
- United States (3):
  - Aurora Clinical Trials, Miami, Florida
  - Community Research, Cincinnati, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
- India (24):
  - Sravani Poly Clinic and Mental Health, Guntur, Andhra Pradesh
  - Asha Hospital, Hyderabaad, Andhra Pradesh
  - Brain Mind Behaviour Neuroscience Research Institute, Maharanipet, Andhra Pradesh
  - VIMHANS, Vijaywada, Andhra Pradesh
  - Government Hospital for Mental Care, Dept. of Psychiatry, Visakhapatnam, Andhra Pradesh
  - SV Medical College, Tirupati, Chittoor District, Andhra Pradesh
  - AIIMS, New Dehli, Dehli
  - Sri Kishna Prasad Psychiatric Nursing Home, Ahmedabad, Gujarat
  - Victoria Hospital, Dept. of Psychiatry, Bangalore, Karnataka
  - St. John's Hospital, Bangalore, Karnataka
  - Adhit Kiran Neuro Psychiatric Centre, Mangalore, Karnataka
  - JSS Medical College Hospital, Dept. of Psychiatry, Mysore, Karnataka
  - Bhopal Memorial Hospital & Research Centre, Dept. of Psychiatry, Bhopal, Madhya Pradesh
  - Holy Family Hospital, Mumbai, Maharashtra
  - Deenanath Maneshkas Hospital, Pune, Maharashtra
  - Sanjeevan Hospital, Pune, Maharashtra
  - Poona Hospital & Research Centre, Pune, Maharashtra
  - GB pant Hospital, Indraprastha, National Capital Territory of Delhi
  - Bhora Nuro Psychiatric Centre, New Delhi, National Capital Territory of Delhi
  - Gautam Hospital & Research Center, Jaipur, Rajasthan
  - Madras Medical College, Chennai, Tamil Nadu
  - M.S. Chellamuthu Trust & Research Foundation, Madurai, Tamil Nadu
  - Mahendru Psychiatric Centre, Kanpur, Uttar Pradesh
  - C.S.M. Medical University, Department of Psychiatry, Lucknow, Uttar Pradesh

REFERENCES:
- [Derived] Khan SA, Revicki DA, Hassan M, Locklear JC, Friedman LA, Mannix S, Tummala R, Dunbar GC, Eriksson H, Sheehan DV. Assessing the Reliability and Validity of the Sheehan Irritability Scale in Patients With Major Depressive Disorder. J Clin Psychiatry. 2016 Aug;77(8):1080-6. doi: 10.4088/JCP.14m09719. PMID 26579723
- [Derived] Xu H, Henningsson A, Alverlind S, Tummala R, Toler S, Beaver JS, Al-Huniti N. Population pharmacokinetics of TC-5214, a nicotinic channel modulator, in phase I and II clinical studies. J Clin Pharmacol. 2014 Jun;54(6):707-18. doi: 10.1002/jcph.264. Epub 2014 Jan 16. PMID 24408516